CLINICAL TRIAL: NCT00218959
Title: Randomized Controlled Trial of Narrative Exposure Therapy Compared to Treatment as Usual for Traumatized Refugees and Asylum Seekers in Mid-Norway
Brief Title: Randomized Controlled Trial of Narrative Exposure Therapy Compared to Treatment as Usual for Traumatized Refugees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Vivo international e.V. (Industry); University of Konstanz (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4.2005.1100
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; trauma treatment; refugees; randomized controlled
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Narrative Exposure Therapy (Experimental): carried out according to the manual as outlined by Schauer et al. (2005) (second revised edition 2011) 10 sessions of 90 min duration
  Interventions: Behavioral: Narrative Exposure Therapy
- treatment as usual (Active Comparator): mainly help with such as sleep problems, depressive symptoms, problems related to asylum status, and other practical matters. Focus on everyday issues and the limited focus on the traumatic events, in line with reports from the National Center on Violence and Traumatic Stress.
  Interventions: Behavioral: treatment as usual

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy — Exposure based treatment for PTSD developed especially for refugees. Built upon Prolonged exposure treatment (Edna Foa) and Testimonial Therapy (Cientifuegos & Monelli).
  Arms: Narrative Exposure Therapy
Behavioral: treatment as usual
  Arms: treatment as usual

SUMMARY:
In this study we want to compare Narrative Exposure Therapy to Treatment as Usual for traumatized refugees and asylum seekers in the Mid- Norway region. Clinicians in psychiatric outpatient clinics will deliver the two conditions to asylum seekers and refugees that qualifies for Posttraumatic Stress Disorder. We will investigate if refugees and asylum seekers will improve more with Narrative Exposure Therapy or Treatment as Usual, and if there will be any differences between improvement for asylum seekers compared to improvement for refugees with residential status.

DETAILED DESCRIPTION:
Narrative Exposure Therapy (NET) will in a randomized controlled trial be compared to Treatment as Usual(TAU) for traumatized refugees and asylum seekers in the Mid- Norway region. Clinicians in psychiatric outpatient clinics in the region will deliver the two conditions to asylum seekers and refugees that qualifies for Posttraumatic Stress Disorder. Each patient will receive 10 sessions of either NET or TAU. Assessment tools in the study will be MINI International Neuropsychiatric Interview, Clinician Administered PTSD Scale and the Hamilton Rating Scale for Depression. Exclusion criteria will be psychosis, substance abuse and serious suicidal ideations. The age group in focus will be adults of 18 years or more. Refugees and asylum seekers from all countries will be accepted in the study, and there will be used qualified interpreters if the refugees do not speak English or Norwegian fluently.

ELIGIBILITY:
Inclusion Criteria:

* Refugee or asylum seeker
* Posttraumatic Stress Disorder diagnosis according to the DSM-IV criteria

Exclusion Criteria:

* Psychosis
* Substance abuse
* Serious suicidal ideations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2005-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale | before treatment, 1 month after, 6 months after

SECONDARY OUTCOMES:
Hamilton Rating Scale for Depression (HAM-D) | before treatment, 1 month after, 6 months after

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Gotestam, Phd, Study Chair — Psychiatric Intitute, NTNU
Locations (1):
- Centre on violence, traumatic stress and suicide prevention - Mid Norway, Trondheim, Trondheim, Norway

REFERENCES:
- [Result] Stenmark H, Catani C, Neuner F, Elbert T, Holen A. Treating PTSD in refugees and asylum seekers within the general health care system. A randomized controlled multicenter study. Behav Res Ther. 2013 Oct;51(10):641-7. doi: 10.1016/j.brat.2013.07.002. Epub 2013 Jul 8. PMID 23916633
- [Derived] Halvorsen JO, Stenmark H, Neuner F, Nordahl HM. Does dissociation moderate treatment outcomes of narrative exposure therapy for PTSD? A secondary analysis from a randomized controlled clinical trial. Behav Res Ther. 2014 Jun;57:21-8. doi: 10.1016/j.brat.2014.03.010. Epub 2014 Apr 12. PMID 24762779
- See also: The developers of Narrative Exposure Therapy — http://www.vivo.org